CLINICAL TRIAL: NCT06596460
Title: Single Centre Prospective Study to Obtain Data to Train an Algorithm for Prediction of Outcome in Transcatheter Aortic Valve Implantation (TAVI)
Brief Title: A Study to Obtain Imaging Data in 40 Patients Having Transcatheter Aortic Valve Implantation (TAVI)
Acronym: CONTINUUM-CT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 164073
Record Dates: First submitted 2024-08-22; First posted 2024-09-19 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Aortic Stenosis, Severe; Aortic Valve Stenosis
Keywords: Heart; Valve; Implantation; Transcatheter; CT; Computerised Tomography
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Acclimatization

STUDY DESIGN:
Intervention Model Description: A single centre, prospective, interventional study in 40 patients undergoing TAVI in a National Health Service (NHS) hospital
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Computerised Tomography (CT) Intervention (Experimental): Transpercutaneous Aortic Valve Implantation (TAVI) planning CT (adapted) of the heart and aortic arch at 6 months post TAVI
  Interventions: Diagnostic Test: TAVI planning CT (adapted)

INTERVENTIONS:
Diagnostic Test: TAVI planning CT (adapted) — TAVI planning CT (adapted) to obtain a standard assessment of the Left Ventricular Outflow Tract (LVOT), valve annulus, aortic root, and ascending aorta up to neck branches. There will be no requirement to scan the ilio-femoral arteries as per standard TAVI planning CT

SUMMARY:
The aim of this study is to learn if the Computed Tomography scan (CT scan) and heart echo scan TransThoracic Echo scan (TTE or heart echo scan) taken before a Transcatheter Aortic Valve Implantation (TAVI) procedure can be used to predict how the new TAVI valve will perform in the future.

To do this the investigators need the usual CT scan before and a new CT scan after the TAVI valve has been put in. At present a CT scan after TAVI procedure is not routinely done. Male and female patients with severe Aortic Stenosis (AS) will be asked to take part.

The data from the scans along with routine measures that are taken will be used to assess if there has been any deterioration in the valve at six months.

The scan data collected will be used in a computer programme. This programme will be trained to predict TAVI valve performance.

The main purpose of this study is to collect the CT scan data before and after the TAVI procedure.

The study aims to answer:

• Can the investigators obtain additional CT imaging data and other data before and after TAVI to enable the prediction of valve performance?

Participants will be asked if they would have another CT scan 6 months after their TAVI procedure, during their routine follow up.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Symptomatic, degenerative, tricuspid, severe aortic stenosis
* TTE derived aortic valve area (AVA) of ≤ 1.0 cm2 (or indexed effective orifice area (EOAi) ≤ 0.6 cm2 /m2)
* TTE derived AV mean gradient ≥ 40 mmHg or peak jet velocity ≥ 4.0 m/s or Doppler Velocity Index (DVI) ≤ 0.25
* CT TAVI deemed of good quality (as per standard operating procedure) within past 6 months
* TTE of good quality within past 6 months as defined by:

  * Doppler signal across the aortic valve and LVOT is a clear and artifact-free waveform
  * Correct alignment to the blood flow direction to ensure accurate velocity measurements
  * Following measurements available
  * Continuous-wave Doppler (CW) across the aortic valve
  * AV Vmax, AV Vmean, AV peak gradient (MaxPG), AV mean gradient (meanPG), AV Velocity-Time integral (VTI), heart rate (HR);
  * Pulse-wave Doppler (PW) across the LVOT
  * LVOT Vmax, LVOT Vmean, LVOT MaxPG, LVOT meanPG, LVOT VTI;
  * 2D LVOT diameter in plax view.
* In sinus rhythm at time of any TTE or CT scans
* Undergone a technically successful elective TAVI as defined by the operator using a Edwards Sapien 3 Ultra (20, 23, 26 or 29 mm):

  * Position and height as planned
  * Trivial aortic regurgitation
  * No vascular or other complications prolonging discharge

Exclusion Criteria:

* Life expectancy <6 months
* Rockwood frailty score >6
* Mixed aortic valve disease with predominant aortic regurgitation that is at least moderate.
* Moderate-severe mitral regurgitation and/or mitral stenosis.
* Congenital unicuspid or congenital bicuspid aortic valve as verified by echocardiography or CT
* Previous TAVI or Aortic Valve Replacement (AVR)
* Left Ventricular Ejection Fraction (LVEF) < 50%
* On or planned oral anticoagulation
* Chronic severe renal failure (estimated glomerule filtration rate (eGFR)) less than 30 mL/min/1.73m2 by the MDRD equation or requiring dialysis)
* Evidence of an acute myocardial infarction within 30 days prior to index procedure
* Untreated clinically significant coronary artery disease requiring revascularization
* Blood dyscrasias as defined: leukopenia (WBC < 3000mm3), acute anaemia (Hb < 9g/dL), thrombocytopenia (platelet count < 50,000 cells/mm3); history of bleeding diathesis or coagulopathy
* Active peptic ulcer or upper GI bleeding within 3 months prior to index procedure that would preclude anticoagulation
* Those lacking capacity to consent or are deemed vulnerable adults
* Requires permanent pacemaker
* Pregnancy or the possibility of pregnancy as reported by the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2026-09-12 (Estimated); Study Completion 2026-09-12 (Estimated)

PRIMARY OUTCOMES:
The number of participants with quality TAVI CT imaging data post TAVI procedure. | At 6 months
  Quality (high-good resolution and without artifacts) retrospectively ECG-gated scan of the heart, aortic annulus and ascending aorta to the first branch vessel. The full body angiogram, best systole and best diastole must be present.

SECONDARY OUTCOMES:
The occurrence of Patient/Prosthesis mismatch (PPM) - as measured by a transvalvular gradient >10 mmHg | At Day 1 post TAVI
The occurrence of haemodynamic valve deterioration as measured by Transthoracic echocardiography (TTE) | At Day 1 post TAVI and 6 months
  Routine measures of Transthoracic echocardiography (TTE) to determine the occurrence of haemodynamic valve deterioration as defined by Valve Academic Research Consortium (VARC -3) criteria
The occurrence of hypo attenuated leaflet thickening (HALT) as reported by radiologist utilising CT scan | At 6 months
Change in New York Heart Association (NYHA) class score I to IV | At baseline and at 6 months
  NYHA functional classification of heart failure classes I to IV where I is best and IV is worst
The occurrence of major adverse cardiac events (MACE) (defined as: cardiovascular death, stroke, myocardial infarction and cardiac reintervention [including stent insertion]) | At 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Mathur, Prof, Principal Investigator — Queen Mary University of London
Locations (1):
- St Bartholomew's Hospital, London, England, United Kingdom